CLINICAL TRIAL: NCT01520818
Title: A Multinational, Randomised, Open-labelled, Parallel Group Four Months Comparison of Twice Daily Biphasic Human Insulin 30 and Thrice Daily Biphasic Insulin Aspart 50 and 70 in Subjects With Type 1 or Type 2 Diabetes
Brief Title: Comparison of Biphasic Human Insulin 30 With Biphasic Insulin Aspart in Subjects With Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-1075
Record Dates: First submitted 2012-01-25; First posted 2012-01-30 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70; biphasic human insulin 30

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BIAsp 50 or 70 (Experimental)
  Interventions: Drug: biphasic insulin aspart 50; Drug: biphasic insulin aspart 70
- BHI 30 (Active Comparator)
  Interventions: Drug: biphasic human insulin 30

INTERVENTIONS:
Drug: biphasic insulin aspart 50 — Administered subcutaneously (s.c., under the skin) at breakfast, lunch and dinner. Randomised subjects being obese with a body mass index (BMI) exceeding 30 kg/m^2 will receive BIAsp 50
  Arms: BIAsp 50 or 70
Drug: biphasic insulin aspart 70 — Administered subcutaneously (s.c., under the skin) at breakfast, lunch and dinner. Randomised subjects being lean and overweight with a body mass index (BMI) of maximum 30 kg/m^2 will receive BIAsp 70
  Arms: BIAsp 50 or 70
Drug: biphasic human insulin 30 — Administered subcutaneously (s.c., under the skin), twice a day
  Arms: BHI 30

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to compare the glycaemic control of biphasic insulin aspart (BIAsp) 70 and/or BIAsp 50 with biphasic human insulin (BHI) 30 treatment.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or Type 2 diabetes
* Current treatment with BHI 30 twice daily as the only insulin therapy for at least 3 months, with or without combination with oral hypoglycaemic agents
* Body mass index (BMI) maximum 40.0 kg/m^2

Exclusion Criteria:

* History of drug or alcohol dependence
* Impaired hepatic function
* Impaired renal function
* Cardiac disease
* Proliferative retinopathy
* Total daily insulin dose at least 1.80 IU/kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 666 (Actual)
Dates: Start 2000-03; Primary Completion 2001-04 (Actual); Study Completion 2001-04 (Actual)

PRIMARY OUTCOMES:
HbA1c (glycosylated haemoglobin A1c)

SECONDARY OUTCOMES:
Blood glucose profiles
Adverse events
Hypoglycaemic episodes
Quality of Life (QoL) assessed via World Health Organization Diabetes Treatment Satisfaction Questionnaire (WHO DTSQ)
Quality of Life (QoL) assessed via Diabetes Health Profile (DHP-2)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR,1452), Study Director — Novo Nordisk A/S
Locations (70):
- Belgium (6):
  - Novo Nordisk Investigational Site, Aalst
  - Novo Nordisk Investigational Site, Brussels
  - Novo Nordisk Investigational Site, Edegem
  - Novo Nordisk Investigational Site, Genk
  - Novo Nordisk Investigational Site, Jumet
  - Novo Nordisk Investigational Site, Liège
- France (26):
  - Novo Nordisk Investigational Site, Amiens
  - Novo Nordisk Investigational Site, Avignon
  - Novo Nordisk Investigational Site, Bagnols-sur-Cèze
  - Novo Nordisk Investigational Site, Bordeaux
  - Novo Nordisk Investigational Site, Caen
  - Novo Nordisk Investigational Site, Colmar
  - Novo Nordisk Investigational Site, Dijon
  - Novo Nordisk Investigational Site, Dommartin-lès-Toul
  - Novo Nordisk Investigational Site, Grenoble
  - Novo Nordisk Investigational Site, La Rochelle
  - Novo Nordisk Investigational Site, Le Creusot
  - Novo Nordisk Investigational Site, Lorient
  - Novo Nordisk Investigational Site, Lyon
  - Novo Nordisk Investigational Site, Marseille
  - Novo Nordisk Investigational Site, Mâcon
  - Novo Nordisk Investigational Site, Nanterre
  - Novo Nordisk Investigational Site, Narbonne
  - Novo Nordisk Investigational Site, Nevers
  - Novo Nordisk Investigational Site, Nîmes
  - Novo Nordisk Investigational Site, Orléans
  - Novo Nordisk Investigational Site, Paris
  - Novo Nordisk Investigational Site, Reims
  - Novo Nordisk Investigational Site, Roubaix
  - Novo Nordisk Investigational Site, Saint-Etienne
  - Novo Nordisk Investigational Site, Strasbourg
  - Novo Nordisk Investigational Site, Toulouse
- Novo Nordisk Investigational Site, Dublin, Ireland
- Netherlands (10):
  - Novo Nordisk Investigational Site, 's-Hertogenbosch
  - Novo Nordisk Investigational Site, Alkmaar
  - Novo Nordisk Investigational Site, Amersfoort
  - Novo Nordisk Investigational Site, Arnhem
  - Novo Nordisk Investigational Site, Beverwijk
  - Novo Nordisk Investigational Site, Delft
  - Novo Nordisk Investigational Site, Einhoven
  - Novo Nordisk Investigational Site, Hengelo
  - Novo Nordisk Investigational Site, Rotterdam
  - Novo Nordisk Investigational Site, The Hague
- United Kingdom (27):
  - Novo Nordisk Investigational Site, Ayr
  - Novo Nordisk Investigational Site, Ayrsh
  - Novo Nordisk Investigational Site, Bath
  - Novo Nordisk Investigational Site, Birmingham
  - Novo Nordisk Investigational Site, Brighton
  - Novo Nordisk Investigational Site, Coventry
  - Novo Nordisk Investigational Site, Dundee
  - Novo Nordisk Investigational Site, Edgware
  - Novo Nordisk Investigational Site, Edinburgh
  - Novo Nordisk Investigational Site, Exeter
  - Novo Nordisk Investigational Site, Glasgow
  - Novo Nordisk Investigational Site, Haywards Heath
  - Novo Nordisk Investigational Site, Ipswich
  - Novo Nordisk Investigational Site, Leeds
  - Novo Nordisk Investigational Site, Leicester
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Manchester
  - Novo Nordisk Investigational Site, Nottingham
  - Novo Nordisk Investigational Site, Paisley
  - Novo Nordisk Investigational Site, Poole
  - Novo Nordisk Investigational Site, Rugby
  - Novo Nordisk Investigational Site, Scunthorpe
  - Novo Nordisk Investigational Site, Southampton
  - Novo Nordisk Investigational Site, Sunderland
  - Novo Nordisk Investigational Site, Swansea
  - Novo Nordisk Investigational Site, Watford
  - Novo Nordisk Investigational Site, Whiston

REFERENCES:
- [Result] Clements MR, Tits J, Kinsley BT, Rastam J, Friberg HH, Ligthelm RJ. Improved glycaemic control of thrice-daily biphasic insulin aspart compared with twice-daily biphasic human insulin; a randomized, open-label trial in patients with type 1 or type 2 diabetes. Diabetes Obes Metab. 2008 Mar;10(3):229-37. doi: 10.1111/j.1463-1326.2006.00687.x. PMID 18269638
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com